CLINICAL TRIAL: NCT06202586
Title: Effect of Different Oxygen Concentration on Postoperative Pulmonary Complications After Pulmonary Reexpansion Following One-lung Ventilation in Thoracic Surgery（DOC-PCT Trial）- A Prospective Randomized Controlled Clinical Study.
Brief Title: Effect of Different Oxygen Concentration on Postoperative Pulmonary Complications After Pulmonary Reexpansion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: The DOC-PCT trial
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Disease
Keywords: postoperative pulmonary complications; thoracic surgery; inspiratory oxygen fraction
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Received low FiO2 (Experimental): Patients undergoing elective thoracic surgery were treated with 30% FiO2 after pulmonary reexpansion following one-lung ventilation and 2-hour postoperative.
  Interventions: Procedure: low FiO2
- Received high FiO2 (Active Comparator): Patients undergoing elective thoracic surgery were treated with 80% FiO2 after pulmonary reexpansion following one-lung ventilation and 2-hour postoperative.
  Interventions: Procedure: high FiO2

INTERVENTIONS:
Procedure: low FiO2 — FiO2 was 100% in two-lung ventilation during anesthesia induction and one-lung ventilation stage intraoperative. FiO2 was 30% in two-lung ventilation after pulmonary reexpansion. During 2 hours after extubation, oxygen was administered through a non-reabsorption mask (high concentration oxygen mask; Intersurgical Ltd, Wokingham, UK) with a respiratory sac in the post anesthesia care unit (PACU), FiO2 was 30% (2L oxygen +14L air per minute). If the subjects who need to be admitted to the intensive care unit (ICU) fail to resuscitate the extubation within a short time after surgery due to their condition and require prolonged respiratory support, FiO2 should be adjusted to 30% 2 hours after admission to the ICU, and respiratory support according to the routine ventilation strategy of ICU should be provided 2 hours later.
  Arms: Received low FiO2
Procedure: high FiO2 — FiO2 was 100% in two-lung ventilation during anesthesia induction and one-lung ventilation stage intraoperative. FiO2 was 80% in two-lung ventilation after pulmonary reexpansion. During 2 hours after extubation, oxygen was administered through a non-reabsorption mask (high concentration oxygen mask; Intersurgical Ltd, Wokingham, UK) with a respiratory sac in the post anesthesia care unit (PACU), FiO2 was 80% (14L oxygen +2L air per minute). If the subjects who need to be admitted to the intensive care unit (ICU) fail to resuscitate the extubation within a short time after surgery due to their condition and require prolonged respiratory support, FiO2 should be adjusted to 80% 2 hours after admission to the ICU, and respiratory support according to the routine ventilation strategy of ICU should be provided 2 hours later.
  Arms: Received high FiO2

SUMMARY:
To evaluate the effect of 80% inspiratory oxygen fraction (FiO2) and 30% FiO2 on the incidence of pulmonary complications after pulmonary reexpansion following one-lung ventilation and 2-hour postoperative within the first 7 days after thoracic surgery, based on lung protective ventilation strategy.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPCs) account for the highest proportion (about 84%) among all the factors leading to death in thoracic surgery. High FiO2 was used in perioperative period. However, there is increasing evidence that high FiO2 in non-thoracic surgery can increase respiratory related adverse events and even mortality. The guideline also suggests that low FiO2 (30-50%) during surgery while ensuring moderate level of oxygenation would be more beneficial to the prognosis of patients. Whereas, the selection of oxygen concentration in thoracic surgery is still unclear, especially which oxygen concentration ventilation is more beneficial to reduce PPCs after pulmonary reexpansion. Strict randomized controlled clinical studies are urgently needed to verify the differences in the incidence of PPCs in patients with different oxygen concentration ventilation strategies. The study aim is to evaluate the effect of 80% FiO2 and 30% FiO2 on the incidence of pulmonary complications after pulmonary reexpansion following one-lung ventilation and 2-hour postoperative within the first 7 days after thoracic surgery, based on lung protective ventilation strategy, and to provide clinical basis for optimizing perioperative management of thoracic surgery and effectively reducing the occurrence of perioperative pulmonary complications

ELIGIBILITY:
Inclusion Criteria:1. Elective thoracic surgery: lung surgery, esophageal surgery, mediastinal surgery, etc.; 2. One-lung ventilation: double lumen bronchial cannula or occluder is used for isolation of one lung; 3, American Society of Anesthesiology (ASA) grade I ~ III; 4, 18 years ≤ age < 80 years; 5. Estimated operation time ≥2 hours; 6. Agree to participate and sign the informed consent.

Exclusion Criteria:

1. Severe lung infection occurs within 1 month;
2. Coronary heart disease or heart failure occurs within 2 or 3 months;
3. Preoperative oxygen saturation is less than 94%; 4, Need continuous oxygen therapy; 5, BMI>35 kg/m2;

6. Pregnant women; 7. Preoperative Hb<70g/L or haematocrit<30%.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of a composite of postoperative pulmonary complications (PPCs) within the first 7 postoperative days | 7 postoperative days
  The incidence of a composite of PPCs within the first 7 postoperative days evaluated by established criteria

SECONDARY OUTCOMES:
Secondary diagnosis of PPCs | 7 postoperative days
  PPCs were defined by established criteria and included respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, and aspiration pneumonitis
Grading of PPCs | 7 postoperative days
  Grading of PPCs evaluated by Clavien-Dindo classification
Grading of surgical complications | 30 postoperative days
  The surgical complications were classified with the Clavien-Dindo classification from grade 0 (no complication) to grade V (death)
Extubation time | immediately after surgery
  The time from the end of surgery to extubation was calculated
Oxygenation index | after extubation and 1 day after surgery
  The oxygenation index after extubation and 1 day after surgery was recorded
Length of stay in ICU | immediately after surgery
  Length of stay in ICU (patients admitted to ICU due to bed turnover are not counted)
Duration of hospitalization | immediately after admission
  Duration of hospitalization were recorded
Incidence of respiratory system related symptoms | 30 postoperative days
  Incidence of respiratory system related symptoms within 30 days after surgery was calculated
All-cause mortality | 30 postoperative days
  All-cause mortality within 30 days after surgery was calculated
PPCs related mortality | 30 postoperative days
  PPCs related mortality within 30 days after surgery was calculated

CONTACTS AND LOCATIONS:
Overall Officials: Wang Xiaojing, M.D., Study Director — Department of Anesthesiology, Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China